CLINICAL TRIAL: NCT04301037
Title: Tension Band Wiring Versus Cannulated Screws in Fixation of Medial Malleolus in Ankle Fracture: Randomized Comparative Study
Brief Title: Tension Band Wiring Versus Cannulated Screws in Fixation of Medial Malleolus in Ankle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU-Sherwan7
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Medial Malleolus Fracture
Keywords: Fixation of medial malleolus; Tension band; Malleolus fracture; Ankle fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tension band wiring (Active Comparator): This group was treated by k-wires fixation and tension band wiring
  Interventions: Procedure: Tension band wires
- Cannulated screws (Active Comparator): This group was treated by 2 cannulated screws
  Interventions: Procedure: Cannulated screws

INTERVENTIONS:
Procedure: Tension band wires — medial malleolus fracture fixed with tension band wiring): 2 k.wires (1.6 mm) are inserted perpendicular to the fracture site. Again the position is checked under image intensification for the correct direction and length. We drilled a 2.5mm hole with a protection sleeve, 2-3cm above the level of the horizontal joint line, aiming the drill bit slightly inferiorly to avoid screw pullout. We inserted a 3.5mm unicortical screw about 30 mm in length (with or without washer), 2-3mm is left for the wire between the bone and screw head before full tightening. A steel wire is constructed into a figure of eight between the screw the reduction k. wires, then twisted to achieve interfragmentary compression
  Arms: Tension band wiring
Procedure: Cannulated screws — In group 2 (15 patients with medial malleolus fixed by 2 cannulated screws): Two guide wires (1.6mm) are inserted perpendicular to the fracture site, the appropriate length, proper insertion site including the distance from the articular surface is checked fluoroscopically .the length is measured .drilling of the bone through the threaded guide wire with a cannulated drill bit (3.2mm). A two 4.5mm partially threaded cannulated screws (with or two washers) are inserted through the guide to achieve Compression, the guide wires are then removed
  Arms: Cannulated screws

SUMMARY:
This is a prospective randomized study conducted on 30 patients with an age spanning between 20 and 55 years. Half of the sample was treated by tension band wiring for closed medial malleolar fractures, and the other half by two cannulated screws. The patients were assessed at (6w-3months and 6months) for clinical and radiological union and evaluated functionally (12 months) using modified Olerund and Molander scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 20-55 years.
2. Isolated or bimalleolar ankle fractures.
3. Closed fractures.

Exclusion Criteria:

1. Patient with poor bone quality on x ray (radiological osteopenia, thinning of the cortices, loss of trabecular definitions and previous insufficiency fractures)
2. Type D isolated medial malleolus, supination adduction (vertical malleolar) fractures.
3. Comminuted fractures.
4. Skeletally immature patients.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Modified Olerund and Molander scoring system | The functional outcome was measured in all patient 12 months after surgery
  Ankle functional outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Sherwan Hamawandi, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No